CLINICAL TRIAL: NCT05233917
Title: The Precision Nutritional Management for MetS (PNMM)
Brief Title: Effects of Olive Oil and MLCT on Glycolipid Homeostasis in Patients With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Yu Zhang, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCT-Olive and MLCT
Record Dates: First submitted 2021-12-29; First posted 2022-02-10 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-02

CONDITIONS: Hyperlipidaemia; Metabolic Syndrome
Keywords: Olive oil; MLCT oil; plasma metabolome; gut microbiota
MeSH Terms: conditions — Hyperlipidemias; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive oil group (Experimental): Olive oil use，25-30 g per day for six month
  Interventions: Dietary Supplement: Olive oil use
- MLCT oil group (Experimental): MLCT oil use，25-30 g per day for six month
  Interventions: Dietary Supplement: MLCT oil use

INTERVENTIONS:
Dietary Supplement: Olive oil use — Olive oil, 25-30g/d by day for 6 month
  Arms: Olive oil group
Dietary Supplement: MLCT oil use — MLCT oil, 25-30g/d by day for 6 month
  Arms: MLCT oil group

SUMMARY:
The type of cooking oil used is a crucial factor influencing dietary quality. The purpose of this study is to investigate the effects of olive oil and MLCT oil intervention on glucose and lipid homeostasis in patients with MetS.

DETAILED DESCRIPTION:
We conducted a 6-month RCT to evaluate the effects of olive oil and MLCT as cooking oils on glucose and lipid homeostasis in patients with MetS; investigate the changes in lipoprotein subfractions and metabolites using NMR spectroscopy, alongside gut microbiota alterations, to elucidate potential mechanisms; and identify baseline variables associated with the anti-obesity effects of olive oil and MLCT.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for the study were those with a confirmed MetS diagnosis according to the IDF criteria53, aged between 40 and 70, and who reported infrequent consumption of meals outside the home (≤3 times per week)

Exclusion Criteria:

(i) current breastfeeding or pregnancy; (ii) history of cardiovascular disease, including heart disease, coronary artery disease, stroke, cerebral infarction, viral hepatitis (e.g., hepatitis A or B), chronic kidney disease (estimated glomerular filtration rate [GFR] <60 ml/min), or malignancy; (iii) presence of diabetic ketoacidosis or hyperketonemia; (iv) recent alterations in prescribed medication within the previous 6 months; (v) current use of insulin therapy; (vi) consumption of MLCT in the preceding 6 months; (vii) participation in other clinical research studies within the last 6 months; and (viii) premenopausal women

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2023-12-09 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Change in body weight from baseline | 6 month
  The investigators will measure body weight of participants before and after treatment.
Change in triglycerides from baseline | 6 month
  The investigators will measure triglyceride levels in blood samples before and after treatment.
Change in Body fat distribution and muscle conten from baseline | 6 month
  The whole body of the patient was scanned and analyzed by a DXA (Prodigy Primo, Dalex-Ohmeda, Inc., USA) to measure the total and regional body fat mass (FM) and lean mass.

SECONDARY OUTCOMES:
Change in waist circumference from baseline | 6 month
  The investigators will measure waist circumference of participants before and after treatment.
Change in MetS indicators from baseline | 6 month
  The investigators will measure TC, LDL-C, HDL-C, and glucose levels in blood samples and blood pressure before and after treatment.
Change in gut microbiota from baseline | 6 month
  The investigators will collect faeces sample from every participants and 16S rDNA sequencing will be used to analyze the composition of gut microbiota.
Change in blood metabolome | 6 month
  The investigators will collect blood samples from every participant and the high-throughput NMR metabolomics platform will be used to analyze the blood metabolomics profile.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhang, PhD, Principal Investigator — Zhejiang University
Locations (1):
- Lanxi Hospital of Traditional Chinese Medicine, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No